CLINICAL TRIAL: NCT01946854
Title: A Randomized Crossover Trial of Systemic Chemotherapy in Patients With Metastatic Well-Differentiated Mucinous Appendiceal Adenocarcinomas With Pseudomyxoma Peritonei
Brief Title: Crossover Trial of Systemic Chemotherapy in Patients With Metastatic Well-Differentiated Mucinous Appendiceal Adenocarcinomas With Pseudomyxoma Peritonei
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2012-1050; NCI-2015-00850 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Gastrointestinal; Metastatic Well-differentiated Mucinous Appendiceal Adenocarcinomas with Pseudomyxoma Peritonea; Appendiceal cancer; Surgically unresectable; Chemotherapy; Observation; Questionnaires
MeSH Terms: conditions — Gastrointestinal Neoplasms; Appendiceal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation Arm (Other): Patients observed for 6 months, then will receive chemotherapy for 6 months.
  Interventions: Behavioral: Questionnaire
- Chemotherapy Group (Active Comparator): Patients receive chemotherapy for 6 months, then observed for 6 months. The exact type of fluoropyrimidine-based chemotherapy is not mandated and final treatment decisions will be left to the medical oncologist who is administering the chemotherapy. All chemotherapy adjustments will be done by the treating medical oncologist according to standard of care.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Completion of 3 questionnaires at baseline and at final visit about quality of life, and 1 questionnaire about symptoms, diagnosis, treatment, prognosis, and patient's relationship with caregivers. These will take about 35-50 minutes to complete.
  Completion of 3 quality of life questionnaires every 3 months for 1 year.

SUMMARY:
Appendiceal cancer is a rare disease that does not cause many symptoms. As such, doctors are not sure if chemotherapy actually has an effect on the disease. The goal of this clinical research study is to learn more about the effects that chemotherapy may have on appendiceal cancer.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups (cohorts):

* If you are in Cohort A, you will first be observed for 6 months, then you will receive chemotherapy for 6 months.
* If you are in Cohort B, you will first receive chemotherapy for 6 months, then you will be observed for 6 months.

You will have an equal chance of being assigned to either cohort. No matter which cohort you are in, the type of chemotherapy you receive will depend on the standard of care for the disease and what your doctor thinks is in your best interest. You will sign a separate consent form for chemotherapy that explains how the drug is given, as well as its risks and benefits.

Study Visits:

Every 3 months (+/- 2 weeks) for 12 months:

* You will have a physical exam, including measurement of your weight and blood pressure.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will complete the 3 questionnaires about your quality of life.
* You will have an MRI or a CT scan to check the status of the disease.

Length of Stud:

You will be on study for up to 12 months. You will no longer be able to take part in this study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your active participation on the study will be over after the end-of-treatment visit.

End-of-Treatment Visit:

The end-of-treatment visit will be the same as your 4th study visit. Twelve (12) months (+/- 4 weeks) after you began the study, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and blood pressure.
* Your performance status will be recorded.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* You will complete the questionnaires you completed at screening.
* If one was not performed within 4 weeks before this visit, you will have an MRI or a CT scan to check the status of the disease.

Long-Term Follow-Up:

After the end-of-treatment visit, you will be followed 1 time each year by checking your medical record and seeing how you are doing. If nothing is in your medical record, you will be called and asked about how you are doing. This call should last about 5-10 minutes.

This is an investigational study.

Up to 30 patients take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histological evidence of a metastatic well differentiated or moderately differentiated mucinous appendiceal epithelial neoplasm (AEN).
2. Radiographic images demonstrating the presence of mucinous peritoneal carcinomatosis (PMP).
3. Patients must not be considered a candidate for a complete surgical cytoreductive surgery. This determination will be made through either discussion at MD Anderson peritoneal surface malignancy multidisciplinary review or consultation with MD Anderson peritoneal surgeon.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
5. Age >/= 18 years old.
6. Patients must be able to understand and provide answers to the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30/OV-28 QOL questionnaires in order to participate in the trial.
7. Adequate bone marrow function as evidenced by: Hemoglobin >/= 9.0 g/dl; Platelet >/= 75,000 cells/mm^3; Absolute neutrophil count >/= 1000/mm^3.
8. Women must not be pregnant or lactating. Women of childbearing potential must have a negative Beta-HCG serum pregnancy test and agree to refrain from breast-feeding, as specified in the informed consent given the unknown risk of teratogenicity of agents in the study. Patients of childbearing potential agree to use an effective form of contraception during chemotherapy and for 90 days following the last chemotherapy treatment.
9. Patients must agree to participate and be able to understand and provide informed consent to participate in the trial.

Exclusion Criteria:

1. Concurrent uncontrolled medical illness that is deemed by the investigator to have potential to interfere with the delivery of chemotherapy for a six month time period.
2. Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 30 days of the first scheduled day of protocol treatment.
3. The presence of complete or partial bowel obstruction based upon clinical assessment.
4. Ongoing use of total parental nutrition.
5. The presence of a concurrent non-appendiceal metastatic cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07-16 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Growth Rate | 6 months
  Primary objective is to determine if difference in tumor growth rate for each patient, as measured by mpRECIST, between observation and systemic chemotherapy periods is ≥5%. Growth rate determined as the percent reduction from the start of the period to the 6 month measurement in that period.

CONTACTS AND LOCATIONS:
Overall Officials: Keith F. Fournier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Shen JP, Yousef AM, Zeineddine FA, Zeineddine MA, Tidwell RS, Beaty KA, Scofield LC, Rafeeq S, Hornstein N, Lano E, Eng C, Matamoros A, Foo WC, Uppal A, Scally C, Mansfield P, Taggart M, Raghav KP, Overman MJ, Fournier K. Efficacy of Systemic Chemotherapy in Patients With Low-grade Mucinous Appendiceal Adenocarcinoma: A Randomized Crossover Trial. JAMA Netw Open. 2023 Jun 1;6(6):e2316161. doi: 10.1001/jamanetworkopen.2023.16161. PMID 37261831
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org